CLINICAL TRIAL: NCT03107975
Title: Effect of Intrathecal Transplant of Human Amniotic Epithelial Cells on Children With Spastic Cerebral Palsy
Brief Title: Effect of Human Amniotic Epithelial Cells on Children With Spastic Cerebral Palsy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: The Second Affiliated Hospital of Fujian Medical University (Other)
Collaborators: Shanghai iCELL Biotechnology Co., Ltd, Shanghai, China (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC-CP
Record Dates: First submitted 2017-04-05; First posted 2017-04-11 (Actual); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Spastic Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cell Therapy (Experimental): intrathecal injection of human amniotic epithelial cells
  Interventions: Biological: human amniotic epithelial cells

INTERVENTIONS:
Biological: human amniotic epithelial cells — intrathecal injection of human amniotic epithelial cells

SUMMARY:
This study aimed to evaluate the therapeutic potential of human amniotic epithelial cell (hAEC) transplant in the management of children with spastic cerebral palsy.

DETAILED DESCRIPTION:
Cerebral palsy is one of the most common congenital (existing at or before birth) disorders of childhood.Spastic cerebral palsy causes stiffness and movement difficulties.There is no cure for the disease now.

This study aimed to evaluate the therapeutic potential of human amniotic epithelial cell (hAEC) transplant in the management of children with spastic cerebral palsy. hAEC will be intrathecal transplanted. Functional status is determined by Gross Motor Function Measure-66 and Fine Motor Function Measure. Spasticity is evaluated by using modified Ashworth scale(MAS).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent document;
* Gross Motor Function Classification System (GMFCS) levels III-V;
* Parents accepted voluntarily cell therapy for their children and followed-up.

Exclusion Criteria:

* Have a history of severe allergic;
* Serological tests such as AIDS, hepatitis B, syphilis, etc;
* Hereditary metabolic diseases of nervous system;
* Tumor or Hematological diseases.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Gross Motor Function Measure-66 | 6 months
  Gross Motor Function Measure-66 is a standardized observational instrument designed and validated to measure change in gross motor function over time in children with cerebral palsy. The scoring key is meant to be a general guideline.

SECONDARY OUTCOMES:
Fine Motor Function Measure | 6 months
  The fine motor performance is evaluated by using Fine Motor Function Measure.
Modified Ashworth Scale | 6 months
  Spasticity is evaluated by using modified Ashworth scale.it is a 6-point scale. Scores range from 0 to 4, where lower scores represent normal muscle tone and higher scores represent spasticity or increased resistance to passive movement.
Gesell Developmental Scales | 6 months
  Neurodevelopmental evaluation with the Gesell Developmental Schedules was performed.

CONTACTS AND LOCATIONS:
Overall Officials: Hongzhi Gao, Dr., Principal Investigator — The Second Affiliated Hospital of Fujian Medical University
Locations (1):
- The Second Affiliated Hospital of Fujian Medical University, Quanzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided